CLINICAL TRIAL: NCT00856297
Title: An Open-Label, Multi-Center Study to Evaluate the Persistence Of Antibody Responses Among Adolescents Who Previously Received Novartis MenACWY Conjugate Vaccine or Commercially Available MenACWY Conjugate Vaccine
Brief Title: Evaluation of Persistence of Anti-meningococcal Bactericidal Antibodies Among Adolescents Who Previously Received MenACWY Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P13E1
Record Dates: First submitted 2009-03-02; First posted 2009-03-05 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Meningococcal Meningitis
Keywords: Meningococcal; ACWY; Conjugate Vaccine; Meningitis; Adolescents; Persistence
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis | interventions — Diphtheria Toxoid

ARMS (5):
- MenACWY-CRM (Experimental): Subjects received one primary dose of MenACWY-CRM conjugate vaccine in the parent study and were followed for persistence in the present study.
  Interventions: Biological: MenACWY-CRM conjugate vaccine
- Licensed comparator (Active Comparator): Subjects received one primary dose of a quadrivalent meningococcal conjugate vaccine with diphtheria toxoid as the protein carrier in the parent study and were followed for persistence in the present study at 5 years postvaccination.
  Interventions: Biological: Licensed comparator
- Naive (Other): Subjects who were age-matched to the other study groups and had not received any previous meningococcal vaccinations.
  Interventions: Biological: MenACWY-CRM conjugate vaccine; Biological: Licensed comparator
- MenACWY-CRM/MenACWY-CRM (Experimental): Subjects received one primary dose of the MenACWY-CRM conjugate vaccine in the parent study and one booster dose of MenACWY-CRM conjugate vaccine at 3 years after primary vaccination.
  Interventions: Biological: MenACWY-CRM conjugate vaccine
- Licensed comparator/MenACWY-CRM (Experimental): Subjects received one primary dose of quadrivalent meningococcal diphtheria toxoid conjugate vaccine in the parent study and one booster dose of MenACWY-CRM conjugate vaccine at 3 years after primary vaccination.
  Interventions: Biological: MenACWY-CRM conjugate vaccine; Biological: Licensed comparator

INTERVENTIONS:
Biological: MenACWY-CRM conjugate vaccine
  Arms: Licensed comparator/MenACWY-CRM; MenACWY-CRM; MenACWY-CRM/MenACWY-CRM; Naive
Biological: Licensed comparator
  Other Names: Quadrivalent meningococcal conjugate vaccine with diphtheria toxoid as the protein carrier
  Arms: Licensed comparator; Licensed comparator/MenACWY-CRM; Naive

SUMMARY:
The primary objective is to evaluate the persistence of bactericidal antibodies in adolescents previously enrolled in the V59P13 study who received either Novartis MenACWY Conjugate Vaccine or commercially available MenACWY conjugate vaccine. The study will also enroll age-matched subjects who have never received any other meningococcal vaccine (naïve subjects) to serve as an additional control group.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in V59P13:

* healthy subjects who have completed the V59P13 study.

Naïve subjects:

* healthy subjects aged-matched with subjects who had completed the V59P13 trial.(currently 16-23 years old).

Exclusion Criteria:

Subjects who had completed the V59P13 study:

* who received any meningococcal vaccine after the V59P13 trial;
* who have had previous confirmed or suspected disease caused by N. meningitidis;
* who have had household contact with and/or intimate exposure to an individual with culture-proven N. meningitidis (serogroups A, C, W135, or Y);
* subjects with any serious, acute or chronic progressive disease.

Naïve subjects:

* who previously received any meningococcal vaccine;
* who have had previous confirmed or suspected disease caused by N. meningitidis;
* who have had household contact with and/or intimate exposure to an individual with culture-proven N. meningitidis (serogroups A, C, W135, or Y);
* subjects with any serious, acute or chronic progressive disease.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 389 (Actual)
Dates: Start 2009-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis
Locations (32):
- United States (32):
  - 37, 50 Birmingham Pediatric Associates 806 Saint Vincent's Drive, Suite 615, Birmingham, Alabama
  - 6 Kaiser Permanente Fremont 39400 Paseo Padre Parkway, Fremont, California
  - 7 Kaiser Permanente Fresno 4785 North First Street, 3rd Floor, Fresno, California
  - 8 Kaiser Permanente Hayward 27303 Sleepy Hollow Ave., 1st Floor, MOB, Hayward, California
  - Admin Kaiser Permanente Vaccine Study Center One Kaiser Plaza, Ordway Building - 16th Floor, Oakland, California
  - 9 Kaiser Permanente Roseville 1840 Sierra Gardens Drive, Vaccine Studies, Roseville, California
  - 11 Kaiser Permanente Sacramento 6600 Bruceville Rd., Pediatric Station C, Sacramento, California
  - Kaiser Permanente, 6600 Bruceville Rd., Sacramento, California
  - 10 Kaiser Permanente San Jose 276 International Circle, Family Health Center, Unit B1, San Jose, California
  - 2 PAMPA 2155 Post Oak Tritt Road, Suite 100, Marietta, Georgia
  - 3 PAMPA 120 Stonebridge Parkway Ste. 410, Woodstock, Georgia
  - 53 Pediatric/Adult Research Inc. 201 South Fifth Street, Suite 102, Bardstown, Kentucky
  - 38 Akron Children's Hospital One Perkins Square, Akron, Ohio
  - 43 Dr. Senders and Associates 2054 South Green Road, South Euclid, Ohio
  - 19 Children's Health Care West 4671 West Lake Road, Erie, Pennsylvania
  - 21 Greenville Medical Centre Inc 90 Shenango Street, Greenville, Pennsylvania
  - 24 (seen at site 21) Family Healthcare Partners 420 Hillcrest Avenue, Grove City, Pennsylvania
  - 23 Pediatric Associates of Latrobe 210 Weldon Street, Latrobe, Pennsylvania
  - 14 Squirrel Hill Office 4070 Beechwood Blvd, Pittsburgh, Pennsylvania
  - 16 Pediatric Alliance Greentree Division 969 Greentree Road Suite 100, Pittsburgh, Pennsylvania
  - 15 South Hills Pediatrics 4411 Stilley Road, Pittsburgh, Pennsylvania
  - 13 Pediatric Alliance Southwestern 850 Clairton Blvd., Pittsburgh, Pennsylvania
  - 20 Pediatric Alliance Arcadia Division 9000 Perry Highway Suite 120, Pittsburgh, Pennsylvania
  - 12 & 18 Primary Physicians Research, Inc. 1580 McLaughlin Run Road, Pittsburgh, Pennsylvania
  - Admin Primary Physicians Research, Inc. 1580 McLaughlin Run Road, Pittsburgh, Pennsylvania
  - 35 Pennridge Pediatric Associates 711 Lawn Avenue, Sellersville, Pennsylvania
  - 22 Laurel Pediatrics 140 Wayland Smith Drive, Uniontown, Pennsylvania
  - 25 Family Practice Medical Associates South 2581 Washington Road Suite 211, Upper Saint Clair, Pennsylvania
  - PEAK Research, LLC, 2589 Washington Road, Suite 412B, Upper Saint Clair, Pennsylvania
  - 47 UTMB Galveston Office of Pediatric Clinical Trials Children's Hospital 301 University Blvd., Rm 1 288H, Galveston, Texas
  - 56 J. Lewis Research, Inc/Foothill Family Clinic South 6360 South 3000 East, Suite 100, Salt Lake City, Utah
  - 45 Group Health Research Institute 1730 Minor Ave, Suite 1600, Seattle, Washington

REFERENCES:
- [Result] Gill CJ, Baxter R, Anemona A, Ciavarro G, Dull P. Persistence of immune responses after a single dose of Novartis meningococcal serogroup A, C, W-135 and Y CRM-197 conjugate vaccine (Menveo(R)) or Menactra(R) among healthy adolescents. Hum Vaccin. 2010 Nov;6(11):881-7. doi: 10.4161/hv.6.11.12849. Epub 2010 Nov 1. PMID 21339701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 19 sites in US.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- Licensed Comparator /MenACWY-CRM: Subjects received one primary dose of quadrivalent meningococcal diphtheria toxoid conjugate vaccine in the parent study and one booster dose of MenACWY-CRM conjugate vaccine at 3 years after primary vaccination.
Period: Overall Study
Arm/Group | MenACWY-CRM | Licensed Comparator | Naive | MenACWY-CRM/MenACWY-CRM | Licensed Comparator /MenACWY-CRM
Started | 131 | 76 | 107 | 44 | 31
Completed | 129 | 76 | 107 | 44 | 31
Not Completed | 2 | 0 | 0 | 0 | 0
Not completed — Unable to classify | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled population
Groups:
- MenACWY-CRM/MenACWY-CRM: Subjects received one primary dose of quadrivalent meningococcal diphtheria toxoid conjugate vaccine in the parent study and one booster dose of MenACWY-CRM conjugate vaccine in the present study at 3 years after primary vaccination.
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM | Licensed Comparator | Naive | MenACWY-CRM/MenACWY-CRM | Licensed Comparator /MenACWY-CRM | Total
Number analyzed (Participants) | 131 | 76 | 107 | 44 | 31 | 389
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.4 (2.4) | 18.8 (2.4) | 19.3 (2.4) | 19.0 (1.9) | 19.7 (2.3) | 19.2 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 29 | 68 | 21 | 13 | 196
  Male | 66 | 47 | 39 | 23 | 18 | 193

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Human Complement Serum Bactericidal Activity (hSBA) Titers≥ 1:8, After One Dose of Either MenACWY-CRM Conjugate or Licensed Comparator Vaccine
Description: Immune response of one dose of MenACWY-CRM conjugate vaccine compared to that of one dose of licensed comparator vaccine at 21 months, 3 years and 5 years after vaccination, as measured by the percentages of subjects with human complement serum bactericidal activity (hSBA) titers≥ 1:8 directed against N meningitidis serogroups A, C, W and Y.
Time Frame: 21 months, 3 years and 5 years postvaccination
Population: Analysis was done on PP persistence population - subjects who provided one evaluable serum sample at baseline at any visit (21 months, 3 years and 5 years) and had no major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM | Licensed Comparator
Number analyzed (Participants) | 102 | 60
percentages of subjects
  MenA - 21 months | 44 [34 to 54] | 27 [16 to 40]
  3 Years | 37 [28 to 47] | 18 [10 to 30]
  5 Years | 34 [25 to 44] | 37 [25 to 50]
  Men C - 21 Months (N=102, 59) | 61 [51 to 70] | 63 [49 to 75]
  3 Years (N=102, 59) | 68 [58 to 77] | 68 [54 to 79]
  5 Years (N=102, 59) | 64 [54 to 73] | 63 [49 to 75]
  MenW- 21 Months (N=101, 57) | 86 [78 to 92] | 60 [46 to 72]
  3 Years (N=101, 57) | 85 [77 to 91] | 65 [51 to 77]
  5 Years (N=101, 57) | 85 [77 to 91] | 70 [57 to 82]
  MenY- 21 Months | 71 [61 to 79] | 53 [40 to 66]
  Three Years | 69 [59 to 77] | 55 [42 to 68]
  Five Years | 67 [57 to 76] | 55 [42 to 68]

2. Secondary Outcome: Percentages of Subjects With hSBA Titers≥ 1:4, After One Dose of Either MenACWY-CRM Conjugate or Licensed Comparator Vaccine
Description: Immune response of one dose of MenACWY-CRM conjugate vaccine compared to that of one dose of licensed comparator vaccine at 21 months, 3 years and 5 years after vaccination, as measured by the percentages of subjects with hSBA titers≥ 1:4 against N meningitidis serogroups A, C, W and Y.
Time Frame: 21 months, 3 years and 5 years postvaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM | Licensed Comparator
Number analyzed (Participants) | 102 | 60
percentages of subjects
  MenA - 21 Months | 44 [34 to 54] | 32 [20 to 45]
  3 Years | 38 [29 to 48] | 22 [12 to 34]
  5 Years | 37 [28 to 47] | 37 [25 to 50]
  MenC - 21 Months (N=102, 59) | 73 [63 to 81] | 71 [58 to 82]
  3 Years (N= 102, 59) | 79 [70 to 87] | 78 [65 to 88]
  5 Years (N=102, 59) | 72 [62 to 80] | 71 [58 to 82]
  MenW - 21 Months (N=101, 57) | 89 [81 to 94] | 61 [48 to 74]
  3 Years (N=101, 57) | 88 [80 to 94] | 67 [53 to 79]
  5 Years (N=101, 57) | 85 [77 to 91] | 70 [57 to 82]
  MenY - 21 Months | 78 [69 to 86] | 63 [50 to 75]
  Three Years | 76 [67 to 84] | 63 [50 to 75]
  Five Years | 74 [64 to 82] | 63 [50 to 75]

3. Secondary Outcome: hSBA Geometric Mean Titers (GMTs), After One Dose of Either MenACWY-CRM Conjugate or Licensed Comparator Vaccine
Description: Immune response of one dose of MenACWY-CRM conjugate vaccine compared to that of one dose of licensed comparator vaccine at 21 months, 3 years and 5 years after vaccination, as measured by the hSBA Geometric Mean Titers (GMTs) against N meningitidis serogroups A, C, W and Y.
Time Frame: 21 months, 3 years and 5 years postvaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-CRM | Licensed Comparator
Number analyzed (Participants) | 102 | 60
titers
  MenA- 21 Months | 6.46 [4.7 to 8.88] | 4.12 [2.84 to 5.99]
  3 Years | 5.51 [3.89 to 7.81] | 3.69 [2.45 to 5.55]
  5 Years | 4.36 [3.09 to 6.14] | 4.92 [3.29 to 7.37]
  MenC - 21 Months (N=102, 59) | 11 [8.01 to 14] | 7.62 [5.38 to 11]
  3 Years (N=102, 59) | 16 [11 to 26] | 17 [10 to 29]
  5 Years (N=102, 59) | 14 [8.74 to 24] | 20 [11 to 35]
  MenW- 21 Months (N=101, 57) | 18 [14 to 25] | 9.3 [6.59 to 13]
  3 Years (N=101, 57) | 31 [21 to 46] | 17 [11 to 28]
  5 Years (N=101, 57) | 32 [21 to 47] | 19 [12 to 31]
  MenY- 21 Months | 14 [10 to 19] | 6.83 [4.76 to 9.79]
  Three Years | 14 [9.68 to 20] | 7.17 [4.68 to 11]
  Five Years | 13 [8.71 to 20] | 8.11 [4.98 to 13]

4. Secondary Outcome: Percentages of Subjects With No Previous Meningococcal Vaccination With hSBA Titers≥ 1:4 and ≥ 1:8
Description: Immune response of age-matched naive subjects with no previous meningococcal vaccination, as measured by the percentages of subjects with hSBA titers≥ 1:4, and ≥ 1:8 against N meningitidis serogroups A, C, W and Y.
Time Frame: day 1
Population: Analysis was done on PP persistence population - subjects who provided one evaluable serum sample at baseline and had no major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | Naive
Number analyzed (Participants) | 106
percentages of subjects
  Men A - hSBA ≥ 1:4 | 11 [6 to 19]
  Men A-hSBA ≥ 1:8 | 8 [3 to 14]
  MenC- hSBA ≥ 1:4 (N=105) | 51 [41 to 61]
  MenC-hSBA ≥ 1:8 (N=105) | 38 [29 to 48]
  MenW - hSBA ≥ 1:4 (N=105) | 66 [56 to 75]
  MenW-hSBA ≥ 1:8 (N=105) | 66 [56 to 75]
  MenY - hSBA ≥ 1:4 (N=105) | 45 [35 to 55]
  MenY-hSBA ≥ 1:8 (N=105) | 39 [30 to 49]

5. Secondary Outcome: hSBA Geometric Mean Titers (GMT) in Subjects With No Previous Meningococcal Vaccination
Description: Immune response of age-matched subjects with no previous meningococcal vaccination, as measured by hSBA geometric mean titers (GMTs) against N meningitidis serogroups A, C, W and Y.
Time Frame: day 1
Population: Analysis was done on PP persistence population (Naive subjects) - subjects who provided one evaluable serum sample at baseline and had no major protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Naive
Number analyzed (Participants) | 106
titers
  MenA | 2.34 [1.73 to 3.16]
  MenC (N=105) | 4.33 [2.72 to 6.88]
  MenW (N=105) | 18 [12 to 27]
  MenY (N=105) | 5.4 [3.61 to 8.1]

6. Secondary Outcome: Percentages of Subjects With hSBA Titers≥ 1:4 and ≥ 1:8 After a Booster Dose of MenACWY-CRM Conjugate Vaccine
Description: Immune response at one month after one dose of MenACWY-CRM conjugate vaccine in subjects who had previously received one dose of MenACWY-CRM conjugate vaccine or licensed comparator vaccine, as measured by percentages of subjects with hSBA Titers≥ 1:4 and ≥ 1:8 against N meningitidis serogroups A, C, W and Y.
Time Frame: 1 month post booster vaccination
Population: Analysis was done on PP post booster persistence population - subjects who provided one evaluable serum sample at baseline at any visit (3 years and 5 years) and had no major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- Licensed Comparator/MenACWY-CRM: Subjects received one primary dose of a quadrivalent meningococcal conjugate vaccine with diphtheria toxoid as the protein carrier in the parent study, and one booster dose of MenACWY- CRM conjugate vaccine in the present study at 3 years after primary vaccination.
Arm/Group | MenACWY-CRM/MenACWY-CRM | Licensed Comparator/MenACWY-CRM
Number analyzed (Participants) | 42 | 30
percentages of subjects
  MenA hSBA ≥ 1:4 | 100 [92 to 100] | 100 [88 to 100]
  MenC≥ 1:4 | 100 [92 to 100] | 100 [88 to 100]
  MenW ≥ 1:4 (N=41, 29) | 100 [91 to 100] | 100 [88 to 100]
  MenY≥ 1:8 | 100 [92 to 100] | 100 [88 to 100]
  MenA hSBA ≥ 1:8 | 100 [92 to 100] | 100 [88 to 100]
  MenC≥ 1:8 | 100 [92 to 100] | 100 [88 to 100]
  MenW ≥ 1:8 (N=41, 29) | 100 [91 to 100] | 100 [88 to 100]
  MenY≥ 1:4 | 95 [84 to 99] | 93 [78 to 99]

7. Secondary Outcome: Percentages of Subjects With hSBA Titers≥ 1:4 and ≥ 1:8 in Subjects After One Dose of MenACWY-CRM Conjugate Vaccine
Description: Persistence of immune response at two years following administration of one dose of MenACWY-CRM conjugate vaccine in subjects who previously received one dose of either MenACWY-CRM conjugate or licensed comparator vaccine, as measured by hSBA titers≥ 1:4 and ≥ 1:8 against N meningitidis serogroups A, C, W and Y.
Time Frame: 2 years postvaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM/MenACWY-CRM | Licensed Comparator /MenACWY-CRM
Number analyzed (Participants) | 44 | 31
percentages of subjects
  MenA hSBA ≥ 1:4 | 77 [62 to 89] | 87 [70 to 96]
  MenA hSBA ≥ 1:8 | 77 [62 to 89] | 77 [59 to 90]
  MenC hSBA ≥ 1:4 | 95 [85 to 99] | 97 [83 to 100]
  MenC hSBA ≥ 1:8 | 95 [85 to 99] | 87 [70 to 96]
  MenW hSBA ≥ 1:4 | 100 [92 to 100] | 97 [83 to 100]
  MenW hSBA ≥ 1:8 | 100 [92 to 100] | 97 [83 to 100]
  MenY hSBA ≥ 1:4 | 98 [88 to 100] | 94 [79 to 99]
  MenY hSBA ≥ 1:8 | 95 [85 to 99] | 94 [79 to 99]

8. Secondary Outcome: Persistence of hSBA Geometric Mean Titers (GMTs) in Subjects After One Dose of MenACWY-CRM Conjugate Vaccine
Description: Persistence of immune response at two years following administration of one dose of MenACWY-CRM conjugate vaccine in subjects who previously received one dose of either MenACWY-CRM conjugate or licensed comparator vaccine, as measured by hSBA GMTs against N meningitidis serogroups A, C, W and Y.
Time Frame: 2 years postvaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-CRM/MenACWY-CRM | Licensed Comparator /MenACWY-CRM
Number analyzed (Participants) | 44 | 31
titers
  MenA | 21 [11 to 38] | 19 [9.79 to 38]
  MenC | 133 [67 to 261] | 61 [29 to 131]
  MenW | 95 [60 to 151] | 114 [68 to 191]
  MenY | 61 [34 to 109] | 46 [24 to 87]

9. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events
Description: Safety was assessed as the number of subjects who had previously been vaccinated in the parent study with MenACWY-CRM or licensed comparator who reported solicited local and systemic adverse events within 7 days after the administration of a booster dose of MenACWY-CRM conjugate vaccine at 3 year time point.
Time Frame: Day 1 to Day 7
Population: Analysis was done on the solicited safety dataset, i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: subjects
Arm/Group | MenACWY-CRM/MenACWY-CRM | Licensed Comparator /MenACWY-CRM
Number analyzed (Participants) | 83 | 77
subjects
  Any Local | 40 | 40
  Injection site pain | 37 | 37
  Injection site erythema | 6 | 7
  injection site induration | 9 | 4
  Any systemic | 41 | 39
  Chills | 9 | 2
  Nausea | 7 | 8
  Malaise | 4 | 8
  Headache | 20 | 21
  Myalgia | 30 | 26
  Arthralgia | 6 | 7
  Rash | 0 | 0
  Fever ( >= 38C ) | 2 | 0
  Others | 15 | 9
  Stayed home | 2 | 1
  Analgesic Antipyretic | 14 | 9

10. Secondary Outcome: Number of Subjects With New Medical Diagnoses of Chronic Diseases, After One Dose of Either MenACWY-CRM Conjugate Vaccine or Licensed Comparator
Description: Safety was assessed in terms of number of subjects with new diagnoses of chronic diseases, among subjects who had previously received one dose of either MenACWY-CRM conjugate vaccine or licensed comparator vaccine.
Time Frame: Day 1 to 5 years
Population: Analysis was done on safety follow-up population - subjects enrolled at 5 years were included in the safety follow-up for 24 hours after blood draw and for analysis of medical history to identify new onset of chronic diseases.
Measure: Number; unit: subjects
Arm/Group | MenACWY-CRM | Licensed Comparator | MenACWY-CRM/MenACWY-CRM | Licensed Comparator /MenACWY-CRM
Number analyzed (Participants) | 284 | 192 | 83 | 77
subjects
  Circulatory system - 21 months | 1 | 0 | 0 | 0
  3 Years | 0 | 0 | 1 | 0
  5 Years | 0 | 0 | 0 | 0
  Digestive system- 21 months | 4 | 1 | 0 | 0
  Digestive system-21 months through 3 years | 1 | 0 | 2 | 0
  Digestive system-3 years through 5 years | 3 | 1 | 0 | 0
  Congenital anomalies - 21 months | 0 | 0 | 0 | 0
  Congenital anomalies-21 months through 3 years | 0 | 1 | 0 | 0
  Congenital anomalies-3 years through 5 years | 0 | 0 | 0 | 0
  Endocrine,nutritional,metabolic,immunity- 21 month | 2 | 0 | 0 | 0
  Endocrine,nutri,met,immun-21 months through 3years | 0 | 0 | 0 | 0
  Endocrine, nutri,met,immun-3 years through 5 years | 2 | 1 | 0 | 0
  Fact. influ. hlth stat & cont. with hlth ser- 21 M | 0 | 1 | 0 | 0
  21 months through 3 years | 0 | 0 | 1 | 0
  3 years through 5 years | 1 | 0 | 0 | 0
  Mental disorders - 21 Months | 8 | 5 | 0 | 0
  Mental disorders-21 months through 3 years | 10 | 6 | 7 | 4
  Mental disorders-3 years through 5 years | 9 | 5 | 2 | 2
  Musculoskeletal sys & connective tissue- 21 Months | 0 | 0 | 0 | 0
  Musculoskeletal sys&conn.tissue-21mth through 3yrs | 1 | 3 | 0 | 1
  Musculoskeletal sys&conn.tissue-3 yrs through 5yrs | 0 | 0 | 0 | 0
  Nervous system and sense organs - 21 Months | 0 | 2 | 0 | 0
  Nervous sys & sense organs-21 mths through 3 years | 2 | 0 | 1 | 1
  Nervous sys & sense organs-3 years through 5 years | 3 | 0 | 2 | 0
  Pregnancy, childbirth, puerperium - 21 Months | 0 | 0 | 0 | 0
  Pregnancy,childbirth,puerperium-21mths through3yrs | 0 | 0 | 0 | 0
  Pregnancy,childbirth,puerperium-3yrs through 5yrs | 1 | 0 | 0 | 0
  Respiratory system - 21 Months | 7 | 3 | 0 | 0
  Respiratory system-21 months through 3 years | 5 | 1 | 5 | 3
  Respiratory system-3 years through 5 years | 7 | 2 | 1 | 0
  Skin and subcutaneous tissue - 21 Months | 0 | 1 | 0 | 0
  Skin &subcutaneous tissue-21 months through 3years | 1 | 2 | 0 | 1
  Skin &subcutaneous tissue-3 years through 5 years | 2 | 2 | 0 | 0
  Symptoms, signs and ill-defined conditions - 21 M | 0 | 0 | 0 | 0
  Symptoms,signs&ill-defined cond-21mths through3yrs | 2 | 0 | 1 | 1
  Symptoms,signs &ill-defined cond-3yrs through 5yrs | 4 | 3 | 0 | 1
  Genitourinary system - 21 M | 1 | 0 | 0 | 0
  Genitourinary system-21 months through 3 years | 0 | 0 | 0 | 0
  Genitourinary system-3 years through 5 years | 3 | 0 | 1 | 0

11. Secondary Outcome: Number of Subjects Who Reported Medically Attended Adverse Events, After One Dose of Either MenACWY-CRM Conjugate or Licensed Comparator Vaccine
Description: Safety was assessed in terms of number of subjects with medically attended AEs within 28 days after vaccination with one dose of either MenACWY-CRM conjugate or licensed comparator vaccine.
Time Frame: 28 days postvaccination
Population: Analysis was done on safety population - subjects who received vaccination with MenACWY-CRM conjugate vaccine, provided post-baseline safety data and provide safety follow-up information for any period during the 28 day follow-up.
Measure: Number; unit: subjects
Arm/Group | MenACWY-CRM | Licensed Comparator | Naive
Number analyzed (Participants) | 82 | 53 | 81
subjects
  Ear and Labyrinth Disorders- Cerumen Impaction | 0 | 1 | 0
  Gastrointestinal Disorders - Stomatitis | 1 | 0 | 0
  Infections & Infestations - Acarodermatitis | 0 | 0 | 1
  Infections & Infestations -Acute Sinusitis | 1 | 0 | 0
  Infections & Infestations -Chlamydial Infection | 0 | 0 | 1
  Infections & Infestations- Genital Herpes | 0 | 0 | 1
  Infections & Inf-Genitourinary Chlamydia Infection | 1 | 0 | 0
  Infections & Infestations- Herpes Zoster | 0 | 0 | 1
  Infections & Infestations - Oral Herpes | 1 | 0 | 0
  Infections & Infestations - Sinusitis | 0 | 0 | 3
  Infections & Infestations - Urinary Tract Infec | 0 | 0 | 1
  Injury and Poisoning - Arthropod Bite | 0 | 0 | 1
  Investigation - Tuberculin Test | 0 | 0 | 1
  Skin &Subcutaneous Tissue Dis- Dermatitis Contact | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: New medical diagnoses of chronic diseases in subjects who previously received MenACWY-CRM conjugate or Licensed comparator vaccine were collected from day 1 to 5 years. Medically attended AEs were collected within 28 days after vaccination at 5 years.
Description: All SAEs reported during 24 hours from blood draw at the 5-year timepoint were collected.
Arm/Group | MenACWY-CRM | Licensed Comparator | Naive | MenACWY-CRM/MenACWY-CRM | Licensed Comparator /MenACWY-CRM
Serious Adverse Events (participants affected / at risk) | 0/284 | 1/178 | 0/343 | 0/83 | 1/77
Other Adverse Events (participants affected / at risk) | 0/284 | 0/178 | 0/343 | 55/83 | 49/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM (N=284) | Licensed Comparator (N=178) | Naive (N=343) | MenACWY-CRM/MenACWY-CRM (N=83) | Licensed Comparator /MenACWY-CRM (N=77)
Death (General disorders) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM (N=284) | Licensed Comparator (N=178) | Naive (N=343) | MenACWY-CRM/MenACWY-CRM (N=83) | Licensed Comparator /MenACWY-CRM (N=77)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 9 | 8
Chills (General disorders) | 0 | 0 | 0 | 9 | 2
Injection site erythema (General disorders) | 0 | 0 | 0 | 6 | 7
Injection site induration (General disorders) | 0 | 0 | 0 | 9 | 4
Injection site pain (General disorders) | 0 | 0 | 0 | 37 | 37
Malaise (General disorders) | 0 | 0 | 0 | 4 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 30 | 26
Headache (Nervous system disorders) | 0 | 0 | 0 | 21 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.